CLINICAL TRIAL: NCT00234286
Title: Intervention to Improve Care at Life's End in VA Medical Centers
Brief Title: Intervention to Improve Care at Life's End
Acronym: BEACON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 03-126
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Results first posted 2015-04-27 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Death; Pain; Dyspnea
Keywords: Palliative Care; Terminal Care; Hospice Care; Patient Care Planning; Nursing Care Plans; Quality of Health Care; Inpatients; Professional education; Resuscitation orders; Pastoral Care
MeSH Terms: conditions — Death; Pain; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Comfort care education intervention, consisting of intensive, on-site staff training together with an electronic order set for palliative care and educational materials
  Interventions: Behavioral: Comfort care education intervention

INTERVENTIONS:
Behavioral: Comfort care education intervention — Comfort care education intervention, consisting of intensive, on-site staff training together with an electronic order set for palliative care and educational materials

SUMMARY:
The BEACON trial (Best Practices for End-of-Life Care for Our Nations' Veterans) was a six-site implementation study to evaluate a multi-component, education-based intervention to improve the quality of end-of-life care provided in VA Medical Centers.

DETAILED DESCRIPTION:
The BEACON trial (Best Practices for End-of-Life Care for Our Nations' Veterans) was a six-site, real-world implementation trial of a multi-component, education-based intervention to improve the quality of end-of-life care conducted in VA Medical Centers (VAMCs).

The primary aim was to evaluate the effectiveness of a multi-component intervention for improving processes of care provided in the last days of life in VAMCs. The second aim was to conduct after-death interviews with next-of-kin and qualitative analysis of their perceptions of the care provided to the veteran and family.

The multi-component intervention targeted VAMC inpatient providers, including physician, nursing, and ancillary staff. It consisted of preparatory site visits, a staff training program, a newly developed Comfort Care order set decision support tool built into the CPRS, and follow-up consultation. The intervention team travelled to each site to conduct two weeks of comprehensive in-service training. Staff were trained to identify actively-dying patients and implement a set of best practices of traditionally home-based hospice care for dying patients. The team provided assistance with policies, procedures, and skill training needed to implement comfort care interventions. Introduction of the intervention at each VAMC was staggered across time at six-month intervals using a multiple-baseline, stepped wedge design.

Data on processes of end-of-life care (last 7 days) were abstracted from the CPRS medical records of all veterans who died before, during, and after the intervention (January 2005-February 2011). A priori, five processes of care were identified as primary endpoints to indicate quality of end-of-life care: 1) presence of an order for opioid pain medication at time of death; 2) a do-not-resuscitate (DNR) order in place at time of death; 3) location of death; 4) presence of enteral feeding tube or intravenous line at time of death; and 5) physical restraints in place at or near time of death.

In addition, in-depth, face-to-face interviews were conducted with 78 bereaved next-of-kin.

ELIGIBILITY:
Inclusion Criteria:

* Aim 1: Not applicable. Patients were deceased.
* Aim 2: After-death interviews with next of kin: must be willing and able to participate in after-death interview at local VA Medical Center.

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2005-08; Primary Completion 2011-03 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn L Burgio, PhD MA BA, Principal Investigator — Birmingham, Alabama VA Medical Center
Locations (1):
- Birmingham VA Medical Center, Birmingham, Alabama, United States

REFERENCES:
- [Background] Williams BR, Woodby LL, Bailey FA, Burgio KL. Identifying and responding to ethical and methodological issues in after-death interviews with next-of-kin. Death Stud. 2008;32(3):197-236. doi: 10.1080/07481180701881297. PMID 18705168
- [Background] Woodby LL, Williams BR, Wittich AR, Burgio KL. Expanding the notion of researcher distress: the cumulative effects of coding. Qual Health Res. 2011 Jun;21(6):830-8. doi: 10.1177/1049732311402095. Epub 2011 Mar 10. PMID 21393618
- [Result] Bailey FA, Williams BR, Goode PS, Woodby LL, Redden DT, Johnson TM 2nd, Taylor JW, Burgio KL. Opioid pain medication orders and administration in the last days of life. J Pain Symptom Manage. 2012 Nov;44(5):681-91. doi: 10.1016/j.jpainsymman.2011.11.006. Epub 2012 Jul 4. PMID 22765968
- [Result] Bailey FA, Allen RS, Williams BR, Goode PS, Granstaff S, Redden DT, Burgio KL. Do-not-resuscitate orders in the last days of life. J Palliat Med. 2012 Jul;15(7):751-9. doi: 10.1089/jpm.2011.0321. Epub 2012 Apr 26. PMID 22536938
- [Derived] Bickel KE, Kennedy R, Levy C, Burgio KL, Bailey FA. The Relationship of Post-traumatic Stress Disorder to End-of-life Care Received by Dying Veterans: a Secondary Data Analysis. J Gen Intern Med. 2020 Feb;35(2):505-513. doi: 10.1007/s11606-019-05538-x. Epub 2019 Dec 2. PMID 31792872
- [Derived] Riggs JS, Woodby LL, Burgio KL, Bailey FA, Williams BR. "Don't get weak in your compassion": bereaved next of kin's suggestions for improving end-of-life care in Veterans Affairs Medical Centers. J Am Geriatr Soc. 2014 Apr;62(4):642-8. doi: 10.1111/jgs.12764. Epub 2014 Mar 21. PMID 24655157
- [Derived] Bailey FA, Williams BR, Woodby LL, Goode PS, Redden DT, Houston TK, Granstaff US, Johnson TM 2nd, Pennypacker LC, Haddock KS, Painter JM, Spencer JM, Hartney T, Burgio KL. Intervention to improve care at life's end in inpatient settings: the BEACON trial. J Gen Intern Med. 2014 Jun;29(6):836-43. doi: 10.1007/s11606-013-2724-6. PMID 24449032
- See also: Growthhouse website MegaSearch, an international clearing house for high quality educational materials related to hospice and palliative care — http://www.growthhouse.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The BEACON trial implemented an intervention to improve quality of care at end of life. Six Veterans Administration Hospitals received the intervention in a pre-post design. Outcomes were abstracted for 6066 individuals who died either pre or post intervention. 78 next-of-kin were enrolled under protocol to conduct qualitative interviews.
Pre-assignment Details: The BEACON trial implemented an intervention to improve quality of care at end of life. Six Veterans Administration Hospitals received the intervention in a pre-post design. Outcomes were abstracted for 6066 individuals who died either pre or post intervention. 78 next-of-kin were enrolled under protocol to conduct qualitative interviews.
Groups:
- BEACON Intervention: Comfort care education intervention, consisting of intensive, on-site staff training together with an electronic order set for palliative care and educational materials
  Comfort care education intervention: Comfort care education intervention, consisting of intensive, on-site staff training together with an electronic order set for palliative care and educational materials
Period: Overall Study
Arm/Group | BEACON Intervention
Started | 6066 (We reviewed eletronic health records for 6066 deceased individuals within 6 VA Hospitals)
Completed | 6066 (We reviewed eletronic health records for 6066 deceased individuals within 6 VA Hospitals)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Deceased veterans
Groups:
- Arm 1: Comfort care education intervention, consisting of on-site staff training together with an electronic order set for palliative care and educational materials
  Comfort care education intervention: Comfort care education intervention, consisting of on-site staff training together with an electronic order set for palliative care and educational materials
Arm/Group | Arm 1
Number analyzed (Participants) | 6066
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.2 (12.0)
Gender [Number; unit: participants] — The total numbers of participants with gender reported is 5921 which differs from the 6066 participant total previously reported. All outcomes and demogaphics for participants were collected by examination of VA electronic records. Gender could not not identified for 145 participants.
  participants
    Female | 109
    Male | 5812
Race/Ethnicity, Customized [Number; unit: participants] — The total numbers of participants with race/ethnicity reported is 5423 which differs from the 6066 participant total previously reported. All outcomes and demogaphics for participants were collected by examination of VA electronic records. Race/ethnicity could not be identified from electronic records for 643 participants.
  participants
    White | 3528
    Black | 1876
    Hispanic white | 8
    Hispanic black | 2
    Native American | 4
    Asian | 1
    Native Hawaiian/Pacific Islander | 4

OUTCOME MEASURES:

1. Primary Outcome: Presence of Order for Opioid Pain Medication
Description: Presence of order for opioid pain medication at time of death based on abstraction of electronic medical record
Time Frame: Pre and Post Intervention
Measure: Number; unit: participants
Groups:
- Pre-Intervention; Post-Intervention: Comfort care education intervention, consisting of intensive, on-site staff training together with an electronic order set for palliative care and educational materials
  Comfort care education intervention: Comfort care education intervention, consisting of intensive, on-site staff training together with an electronic order set for palliative care and educational materials
Arm/Group | Pre-Intervention | Post-Intervention
Number analyzed (Participants) | 3243 | 2823
participants | 2004 | 2056
Statistical Analysis 1: Comparison: Pre-Intervention vs Post-Intervention; Test type: Superiority or Other; p = .009, Generalized Estimating Equation; Odds Ratio (OR) = 1.39, 95% CI 2-sided [1.09 to 1.76]

2. Secondary Outcome: Do Not Resuscitate Order
Description: Presence of a Do Not Resuscitate order at time of death based on abstraction of electronic medical record
Time Frame: Pre and Post Intervention
Measure: Number; unit: participants
Arm/Group | Pre-Intervention | Post-Intervention
Number analyzed (Participants) | 3243 | 2823
participants | 2282 | 2127
Statistical Analysis 1: Comparison: Pre-Intervention vs Post-Intervention; Test type: Superiority or Other; p = 0.09, Generalized Estimating Equation; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.95 to 1.96]

3. Secondary Outcome: Number of Patients Who Died in ICU
Description: Location of death (ICU vs. other) based on abstraction of electronic medical record
Time Frame: Pre and Post Intervention
Measure: Number; unit: participants
Groups:
- Pre-Intervention: Number of Individuals who died in ICU Pre-Intervention
- Post-Intervention: Number of Patients who died in ICU Post-Intervention
Arm/Group | Pre-Intervention | Post-Intervention
Number analyzed (Participants) | 3243 | 2823
participants | 1312 | 1046
Statistical Analysis 1: Comparison: Pre-Intervention vs Post-Intervention; Test type: Superiority or Other; p = 0.69, Generalized Estimating Equation; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.59 to 1.42]

4. Secondary Outcome: Individuals With a Nasogastric Tube
Description: Presence of nasogastric tube based on abstraction of electronic medical record
Time Frame: Pre and Post Intervention
Measure: Number; unit: participants
Groups:
- Pre-Intervention: Individuals who died with a nasogastric tube pre-intervention
- Post-Intervention: Individuals who died with a nasogastric tube post-intervention
Arm/Group | Pre-Intervention | Post-Intervention
Number analyzed (Participants) | 3243 | 2823
participants | 1293 | 922
Statistical Analysis 1: Comparison: Pre-Intervention vs Post-Intervention; Test type: Superiority or Other; p = .03, Generalized Estimating Equations; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.53 to 0.96]

5. Secondary Outcome: Individuals With an Intravenous Line
Description: Presence of intravenous line infusing at time of death based on abstraction of electronic medical record
Time Frame: Pre and Post Intervention
Measure: Number; unit: participants
Groups:
- Pre-Intervention: Individuals who died with an intravenous line pre-intervention
- Post-Intervention: Individuals who died with an intravenous line post-intervention
Arm/Group | Pre-Intervention | Post-Intervention
Number analyzed (Participants) | 3243 | 2823
participants | 2004 | 2056
Statistical Analysis 1: Comparison: Pre-Intervention vs Post-Intervention; Test type: Superiority or Other; p = 0.15, Generalized Estimating Equation; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.38 to 1.16]

6. Secondary Outcome: Number of Individuals Who Died in Restraints
Description: Presence of restraints at or near time of death at time of death based on abstraction of electronic medical record
Time Frame: Pre and Post Intervention
Measure: Number; unit: participants
Groups:
- Pre-Intervention: Individuals who died with restraints during pre-intervention
- Post-Intervention: Individuals who died with restraints during post-intervention
Arm/Group | Pre-Intervention | Post-Intervention
Number analyzed (Participants) | 3243 | 2823
participants | 531 | 362
Statistical Analysis 1: Comparison: Pre-Intervention vs Post-Intervention; Test type: Superiority or Other; p = 0.86, Generalized Estimating Equation; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.67 to 1.62]

7. Secondary Outcome: Individuals Administered of Opioid Medication
Description: Administration of opioid medication based on abstraction of medical record
Time Frame: Pre and Post Intervention
Measure: Number; unit: participants
Groups:
- Pre-Intervention: Individuals who received opioid medication pre-intervention
- Post-intervention: Individuals who received opioid medication post-intervention
Arm/Group | Pre-Intervention | Post-intervention
Number analyzed (Participants) | 3243 | 2823
participants | 1569 | 1662
Statistical Analysis 1: Comparison: Pre-Intervention vs Post-intervention; Test type: Superiority or Other; p = 0.09, Generalized Estimating Equation; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.95 to 1.96]

8. Secondary Outcome: Individuals With an Order for Antipsychotic Medication
Description: Order for antipsychotic medication based on abstraction of medical record
Time Frame: Pre and Post Intervention
Measure: Number; unit: participants
Groups:
- Pre-Intervention: Individuals with antipsychotic medication ordered pre-intervention
- Post-Intervention: Individuals with antipsychotic medication ordered post-intervention
Arm/Group | Pre-Intervention | Post-Intervention
Number analyzed (Participants) | 3243 | 2823
participants | 336 | 661
Statistical Analysis 1: Comparison: Pre-Intervention vs Post-Intervention; Test type: Superiority or Other; p = 0.01, Generalized Estimating Equation; Odds Ratio (OR) = 1.98, 95% CI 2-sided [1.17 to 3.36]

9. Secondary Outcome: Individuals Administered Antipsychotic Medication
Description: Administration of antipsychotic medication based on abstraction of medical record
Time Frame: Pre and Post Intervention
Measure: Number; unit: participants
Groups:
- Pre-Intervention: Individuals with Administration of antipsychotic medication pre-intervention
- Post-Intervention: Individuals with Administration of antipsychotic medication post-intervention
Arm/Group | Pre-Intervention | Post-Intervention
Number analyzed (Participants) | 3243 | 2823
participants | 224 | 280
Statistical Analysis 1: Comparison: Pre-Intervention vs Post-Intervention; Test type: Superiority or Other; p = 0.36, Generalized Estimating Equation; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.73 to 2.35]

10. Secondary Outcome: Individuals With an Order for Benzodiazepine Medication
Description: Order for benzodiazepine medication based on abstraction of medical record
Time Frame: Pre and Post Intervention
Measure: Number; unit: participants
Groups:
- Pre-Intervention: Individuals with Order for benzodiazepine medication during pre-intervention period based on abstraction of medical record
- Post-Intervention: Individuals with Order for benzodiazepine medication during post-intervention period based on abstraction of medical record
Arm/Group | Pre-Intervention | Post-Intervention
Number analyzed (Participants) | 3243 | 2823
participants | 1102 | 1185
Statistical Analysis 1: Comparison: Pre-Intervention vs Post-Intervention; Test type: Superiority or Other; p = 0.01, Generalized Estimating Equation; Odds Ratio (OR) = 1.39, 95% CI 2-sided [1.08 to 1.77]

11. Secondary Outcome: Individuals Who Received Benzodiazepine Medication
Description: Administration of benzodiazepine medication based on abstraction of medical record
Time Frame: Pre and Post Intervention
Measure: Number; unit: participants
Groups:
- Pre-Intervention: Individuals with Administration of benzodiazepine medication during pre-intervention based on abstraction of medical record
- Post-Intervention: Individuals with Administration of benzodiazepine medication during post-intervention based on abstraction of medical record
Arm/Group | Pre-Intervention | Post-Intervention
Number analyzed (Participants) | 3243 | 2823
participants | 710 | 675
Statistical Analysis 1: Comparison: Pre-Intervention vs Post-Intervention; Test type: Superiority or Other; p = 0.76, Generalized Estimating Equation; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.70 to 1.30]

12. Secondary Outcome: Individuals Who Received Scopolamine
Description: Administration of scopolamine (for death rattle) based on abstraction of medical record
Time Frame: Pre and Post Intervention
Measure: Number; unit: participants
Groups:
- Pre-Intervention: Individuals with Administration of scopolamine (for death rattle) during pre-intervention based on abstraction of medical record
- Post-Intervention: Individuals with Administration of scopolamine (for death rattle) during post -intervention based on abstraction of medical record
Arm/Group | Pre-Intervention | Post-Intervention
Number analyzed (Participants) | 3243 | 2823
participants | 113 | 633
Statistical Analysis 1: Comparison: Pre-Intervention vs Post-Intervention; Test type: Superiority or Other; p = .004, Generalized Estimating Equation; Odds Ratio (OR) = 2.77, 95% CI 2-sided [1.41 to 5.44]

13. Secondary Outcome: Sublingual Administration
Description: Sublingual administration of medication based on abstraction of medical record
Time Frame: Pre and Post Intervention
Measure: Number; unit: participants
Groups:
- Pre-Intervention: Individuals with Sublingual administration of medication during pre-intervention based on abstraction of medical record
- Post-Intervention: Individuals with Sublingual administration of medication during post-intervention based on abstraction of medical record
Arm/Group | Pre-Intervention | Post-Intervention
Number analyzed (Participants) | 3243 | 2823
participants | 122 | 322
Statistical Analysis 1: Comparison: Pre-Intervention vs Post-Intervention; Test type: Superiority or Other; p = 0.007, Generalized Estimating Equations; Odds Ratio (OR) = 4.12, 95% CI 2-sided [1.51 to 11.28]

14. Secondary Outcome: Individuals With Pastoral Care Visit
Description: Pastoral Care Visit based on abstraction of medical record
Time Frame: Pre and Post Intervention
Measure: Number; unit: participants
Groups:
- Pre-Intervention: Individuals with Pastoral Care Visit pre-intervention based on abstraction of medical record
- Post-Intervention: Individuals with Pastoral Care visit post-intervention based on abstraction of medical record
Arm/Group | Pre-Intervention | Post-Intervention
Number analyzed (Participants) | 3243 | 2823
participants | 1630 | 1765
Statistical Analysis 1: Comparison: Pre-Intervention vs Post-Intervention; Test type: Superiority or Other; p = 0.14, Generalized Estimating Equations; Odds Ratio (OR) = 1.64, 95% CI 2-sided [0.84 to 3.20]

15. Secondary Outcome: Individuals With an Advance Directive
Description: Presence of advance directive based on abstraction of medical record
Time Frame: Pre and Post Intervention
Measure: Number; unit: participants
Groups:
- Pre-Intervention: Individuals with Advanced Directive pre-intervention based on abstraction of medical record
- Post-Intervention: Individuals with Advanced Directive post-intervention based on abstraction of medical record
Arm/Group | Pre-Intervention | Post-Intervention
Number analyzed (Participants) | 3243 | 2823
participants | 1194 | 1306
Statistical Analysis 1: Comparison: Pre-Intervention vs Post-Intervention; Test type: Superiority or Other; p = .003, Generalized Estimating Equation; Odds Ratio (OR) = 1.47, 95% CI 2-sided [1.15 to 1.88]

16. Secondary Outcome: Individuals With a Palliative Care Consultation
Description: Palliative Care Consultation based on abstraction of medical record
Time Frame: Pre and Post Intervention
Measure: Number; unit: participants
Groups:
- Pre-Intervention; Post-Intervention: Individuals with documented Palliative Care Consultation pre-intervention in their medical record
Arm/Group | Pre-Intervention | Post-Intervention
Number analyzed (Participants) | 3243 | 2823
participants | 184 | 885
Statistical Analysis 1: Comparison: Pre-Intervention vs Post-Intervention; Test type: Superiority or Other; p = 0.19, Generalized Estimation Equations; Odds Ratio (OR) = 2.45, 95% CI 2-sided [0.62 to 9.70]

ADVERSE EVENTS:
Time Frame: Adverse and Serious Event data were not collected.
Description: All observations were retrospectively collected from electronic records to examine standard of care at the end of life. Therefore, the total number of individuals at risk is 0 because serious and adverse effects were not collected on the 6066 deceased individuals for whom electronic records were abstracted.
Groups:
- Arm 1: Arm 1: Comfort care education intervention, consisting of intensive, on-site staff training
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes